CLINICAL TRIAL: NCT04315259
Title: Efficiency of Diode Laser in Control of Post-endodontic Pain (A Randomized Clinical Trial )
Brief Title: Efficiency of Diode Laser in Control of Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hend Hamdy Ismail, Principle Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: END 16-13D
Record Dates: First submitted 2020-03-07; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Periapical Diseases
Keywords: Diode laser; low laser therapy
MeSH Terms: conditions — Periapical Diseases | interventions — Lasers, Semiconductor; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: study is Single Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laser activated irrigation (Experimental): conventional root canal treatment was done , 2.5% sodium hypochlorite was used and was activated by 980 nm with a repeated pulse mode using a pulse duration of 5 s and a pulse interval of 0.2 ms. The laser irradiation will be delivered for 1 minute into the canal up to 1 mm short of the working length, with circling movements from the apical part moving towards the coronal part (Lite Medics 1.00Watt serial number 148 Ver.SwvM. 150VS108VT.100)
  Interventions: Device: Diode laser
- Soft tissue laser application (Experimental): Endodontically treated teeth by virtue of a dental applicator positioned at a right angle to the mucosa at the level of the apices.
  Application of the laser probe was applied to both the buccal and lingual mucosae overlying the apices of the target tooth. Total exposure time for each tooth was 60 seconds (a dose = 70 j/cm2 for analgesia) The laser unit used in this study used was a diode laser (Lite Medics 1.00Watt serial number 148 Ver.SwvM. 150VS108VT.100) of wavelength 980nm and Max power 15WCW Class IV Laser Product
  Interventions: Device: Diode laser
- conventional root canal (No Intervention): conventional root canal treatment with irrigation of sodium hypochlorite 2.5% with no laser intervention

INTERVENTIONS:
Device: Diode laser — irrigation activated by diode laser versus soft tissue laser application therapy
  Other Names: Low laser therapy; soft laser; Lite medics serial number 148 Ver.SwvM. 150VS108VT.100
  Arms: Laser activated irrigation; Soft tissue laser application

SUMMARY:
Study is a Randomized clinical trial conducted at Endodontic department- Ain Shams university Cairo. Egypt.

180 eligible patients were selected and included in the study to assess the post-endodontic pain of diode laser activated irrigation versus soft tissue diode laser application post obturation versus conventional root canal treatment .

DETAILED DESCRIPTION:
Sample size is 180 180 Patients were randomly distributed in 3 groups , one group of patients received laser therapy after root canal treatment and the other group received disinfection by Diode laser activated irrigation , the third group received no treatment just conventional Root canal treatment. • Patients were equally divided into 3 groups (n=60 in each group ) The study in a Single blinded Randomized clinical trial

, Numbers for patients will be generated and distributed randomly in a table on an Excel sheet, and in front of each number either a letter (C) for control or (I) for intervention will be typed After patients were selected in the study they will be asked to fill in a consent form , that states that they are part of a clinical trial and that they may or may not have a laser session following root canal treatment to test its ability to control pain , the consent will also require them to take a questionnaire at home to measure their pain level and they were willingly do it.

Conventional root canal treatment were done to selected teeth , and any cases with procedural errors were excluded.

Group A Laser activated irrigation :Disinfection were done by using 5 ml of 2.5% sodium hypochlorite irrigation for 1 minute. Irrigation will be performed with a 30-gauge needle side vented The irrigation needles were introduced passively up to 2 mm away the working length. After irrigation Laser treatment will be performed with a diode laser, at a wavelength of 980 nm with a repeated pulse mode using a pulse duration of 5s per canal and a pulse interval of 0.2 ms. The laser irradiation were delivered for 1 minute into the canal up to 1 mm short of the working length, with circling movements from the apical part moving towards the coronal part Group B Soft tissue laser application : Endodontically treated teeth were targeted by virtue of a dental applicator positioned at a right angle to the mucosa at the level of the apices. Application of the laser probe were applied to both the buccal and lingual mucosae overlying the apices of the target tooth. Total exposure time for each tooth was 60 seconds (a dose = 70 j/cm2 for analgesia) by the co-investigator The laser unit used in this study will be a diode laser (Lite Medics 1.00 Watt serial number 148 Ver.SwvM. 150VS108VT.100) of wavelength 980nm and Max power 15 WCW Class IV Laser Product ) in continuous wave mode Group C : conventional root canal treatment : no laser intervention Patients were instructed to record their post-endodontic pain by VAS where 0 stands for no pain and 10 stands for severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age between 18-50 years
* Medically free patients.
* Patients suffering from acute or chronic infection with symptomatic apical periodontitis with Necrotic pulp
* Preoperative Pain
* Sensitivity to percussion
* Periapical radiographic X-ray showing periapical lesion with no gutta percha in canal
* Occlusal contact with opposing teeth

Exclusion Criteria:

* Pregnant females.
* Patients having a significant systemic disorder or history of drug abuse
* Patients who had administrated analgesics or antibiotics during the last 12 hours preoperatively.
* Patients having bruxism or clenching
* Teeth having:

  * No occlusal contact
  * No sensitivity to percussion
  * Greater than grade I mobility.
  * Pocket depth greater than 5mm.
  * No possible restorability
  * Procedural errors
  * Previous Root canal treatment
  * Open apex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Measure change in post-operative pain after Laser intervention using a visual analogue scale (VAS) questionnaire where 0 indicates no pain and 10 indicates severe pain | 24 hours
Measure change in post-operative pain after Laser intervention using a visual analogue scale (VAS) questionnaire where 0 indicates no pain and 10 indicates severe pain | 48 hours
Measure change in post-operative pain after Laser intervention using a visual analogue scale (VAS) questionnaire where 0 indicates no pain and 10 indicates severe pain | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Maram Obeid, PhD, Study Director — Ainshams University; Ehab Hassanien, PhD, Study Chair — Ainshams University
Locations (1):
- Endodontic department - Faculty of Dentistry Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No